CLINICAL TRIAL: NCT06340555
Title: Multiprofessional Healthcare Intervention to Prevent Mental Health Disorders of Women and Their Partners Who Experienced Pregnancy Loss (Enzo Study): A Hybrid Controlled Clinical Trial
Brief Title: Intervention to Prevent Mental Health Disorders of Women and Their Partners Who Experienced Pregnancy Loss
Acronym: Enzo
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: University of Barcelona (Other); University of Seville (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PIC-156-22
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Stillbirth and Fetal Death
MeSH Terms: conditions — Stillbirth; Fetal Death

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enzo intervencion group (Experimental): The hospital 1 guide for care consists on a multidisciplinary team intervention on three moments related to the loss: diagnose, intrapartum, postpartum.
  1. Diagnose: we aim to inform, prepare following procedures and support in the decision-making.
  2. Intrapartum: we aim to reduce or even avoid trauma caused by the situation.
  3. Postpartum: we aim to ensure mother and partner are able to say good-bye absolutely how they planned and/or desire at each time. Also, coordinate continuum of care after hospital discharge.
  Interventions: Other: GUIA ATENCION MULTIDISCIPLINAR SANT BOI
- Control group (Active Comparator): It is the usual care intervention which consists in: diagnosis given by the doctor, intrapartum routine care and follow up on discharge by gynaecologist team.
  Interventions: Other: USUAL CARE

INTERVENTIONS:
Other: GUIA ATENCION MULTIDISCIPLINAR SANT BOI — Women with losses attended according to the multidisciplinary intervention proposed at the SJD Hospital de Sant Boi
  Arms: Enzo intervencion group
Other: USUAL CARE — Women with losses treated at the Hospital Comarcal del l'Alt Penedes.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to test impact of a multiprofessional intervention in mothers and partners who suffer a pregnancy loss. The main questions it aims to answer are:

* impact on mothers and partners mental heatlht status
* reasons why mothers do not consent to the intervention

Participants will:

* mothers and partners will complete 4 scales
* mothers and partners will participate in a interview

Researchers will compare with mothers with standard care to see if the multiprofessional intervention has an impact.

DETAILED DESCRIPTION:
Objective 1: Evaluate the effectiveness of the multi professional intervention to reduce the intensity of grief, depression, anxiety and PTSD symptoms in women and their partners after pregnancy loss.

Objective 2: Assess the extent to which the multiprofessional intervention was implemented as intended (fidelity) and understand how the intervention becomes integrated into routine healthcare practice (implementation).

ELIGIBILITY:
Inclusion Criteria:

* Women and their partners who suffer a pregnancy loss
* Health professionals who have worked for at least 1 year in the hospital studied

Exclusion Criteria:

* Participants who do not understand spanish/catalan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Intensity of grief | 6 months
  Measured with Perinatal Grief Score (PGS Scale)

SECONDARY OUTCOMES:
Depressive symptoms | 6 months
  Measured with Edinburgh Scale
Anxiety symptoms | 6 months
  Measured with Generalized Anxiety Disorder (GAD-7 Scale)
Perinatal postraumatic stress disorder | 6 months
  Measured with Perinatal Postraumatic Questionnaire (PPQ Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Parc Sanitari Sant Joan de Deu, Sant Boi de Llobregat, Barcelona, Spain